CLINICAL TRIAL: NCT03792152
Title: A Prospective Randomized Controlled Trial of Rivaroxaban Versus Warfarin in Dissolving Left Atrial Appendage Thrombus in Patients With Atrial Fibrillation
Brief Title: A Trial of Rivaroxaban Versus Warfarin in Dissolving Left Atrial Appendage Thrombus in Patients With Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, professor, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REVIEW-AF
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Thrombosis; Rivaroxaban
Keywords: Atrial Fibrillation; Left Atrial Appendage Thrombosis; rivaroxaban
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Intervention Model Description: two groups, group one is for Rivaroxaban 20mg qd (15mg qd If creatinine clearance is between 30-49ml/min), group two is for warfarin, keep the INR between 2-3.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After receiving the informed consent form patient, The heads of the centers randomly extracted the envelopes and patients are included in the study based on random envelope grouping results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rivaroxaban (Experimental): After diagnosis of left atrial appendage thrombus by transesophageal echocardiography, then start with rivaroxaba 20mg qd(15mg If creatinine clearance is between 30-49 ml/min ).
  Interventions: Drug: Rivaroxaban
- Warfarin (Active Comparator): After diagnosis of left atrial appendage thrombus by transesophageal echocardiography, subcutaneous injection of low molecular weight heparin and oral warfarin treatment were started, and low molecular weight heparin was stopped after INR reached 2.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — After diagnosis of left atrial appendage thrombus by transesophageal echocardiography, then start with rivaroxaba 20mg qd (15mg If creatinine clearance is between 30-49 ml/min).
  Arms: rivaroxaban
Drug: Warfarin — After the diagnosis of left atrial appendage thrombus by transesophageal echocardiography, subcutaneous injection of low molecular weight heparin (4000iu q12h) and oral warfarin treatment were started, and low molecular weight heparin was stopped after INR reached 2.
  Arms: Warfarin

SUMMARY:
The purpose of this clinical randomized trial is to evaluate the efficacy and safety of rivaroxaban compared with warfarin in dissolving the LAA thrombus in patients with atrial fibrillation.

DETAILED DESCRIPTION:
Left atrial appendage (LAA) thrombosis is a common complication of atrial fibrillation and will significantly increase the incidence of stroke in patients. Warfarin is a classical oral anticoagulant which can dissolve thrombus, but its clinical use has many limitations and it requires strict monitoring of coagulation. Recently, some studies have shown that NOAC (dabigatran / rivaroxaban) can dissolve left atrial appendage thrombosis. The application of rivaroxaban in the X-TRA study dissolved 41.5% of LAA thrombus after 6 weeks, indicating its potential clinical application prospects. Whether rivaroxaban is not inferior to warfarin for rapid dissolution of LAA thrombus, there is no prospective randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Get informed consent from the patient or family.
2. Non-valvular atrial fibrillation / atrial flutter.
3. The first transesophageal echocardiogram revealed a left atrial appendage thrombus (within 7 days of detection of thrombus).
4. Age at 18-80 years old.
5. CrCL≥ 30 mL/min (Cockcroft-Gault).
6. AST/ALT is less than 2 times the upper limit of normal.
7. Women of childbearing age need contraception.

Exclusion Criteria:

1. Pregnant or lactating woman.
2. Can't understand or follow the research plan.
3. Patients under 18 or over 80 years old.
4. Low weight (< 40 kg).
5. Previously found LAA thrombus and have taken anticoagulant drugs.
6. Patients with contraindications for anticoagulation.
7. Patients who need to use antiplatelet drugs simultaneously within 6-12 months after ACS or PCI.
8. A history of cerebral hemorrhage.
9. Patients with active bleeding.
10. Severe gastritis, gastroesophageal reflux patients.
11. Combination of P-glycoprotein inhibitors and other drugs in the presence of NOAC contraindications.

13.Patient with tumor. 14.Planned surgery within 3 months. 15.Other investigators believe that patients are not suitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patient who's thrombus in the left atrium or left atrial appendage is completely dissolved within 3 to 6 weeks | 6 weeks
  Transesophageal echocardiography was used to assess whether there was a left atrial appendage thrombus at 3rd, 6th week after initiation of anticoagulant therapy.

SECONDARY OUTCOMES:
Number of patient who's thrombus in the left atrium or left atrial appendage is completely dissolved within 12 weeks | 12 weeks
  Transesophageal echocardiography was used to assess whether there was a left atrial appendage thrombus at 12th week after initiation of anticoagulant therapy.
Size change of left atrial appendage or left atrium thrombus | 12 weeks
  If a left atrial appendage or left atrial thrombus is detected,then the size of the thrombus is measured using echocardiography。
Number of severe bleeding cases such as gastrointestinal bleeding and cerebral hemorrhage. | 12 weeks
  Number of severe bleeding cases such as gastrointestinal bleeding and cerebral hemorrhage.
Number of transient ischemic attacks (TIA) and strokes | 12 weeks
  Number of transient ischemic attacks (TIA) and strokes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lip GY, Hammerstingl C, Marin F, Cappato R, Meng IL, Kirsch B, van Eickels M, Cohen A; X-TRA study and CLOT-AF registry investigators. Left atrial thrombus resolution in atrial fibrillation or flutter: Results of a prospective study with rivaroxaban (X-TRA) and a retrospective observational registry providing baseline data (CLOT-AF). Am Heart J. 2016 Aug;178:126-34. doi: 10.1016/j.ahj.2016.05.007. Epub 2016 May 17. PMID 27502860